CLINICAL TRIAL: NCT00308061
Title: Double Blind Randomized Controlled Phase I Trial to Evaluate the Safety and Immunogenicity of WRAIR's MSP1 Candidate Malaria Vaccine (FMP1) Adjuvant in GSK Bio's AS02A vs. Rabies Vaccine in Semi-immune Adults in Bandiagara, Mali.
Brief Title: Safety Study of Candidate Malaria Vaccine FMP1/AS02A in Healthy Adults in Bandiagara, Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); GlaxoSmithKline (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRAIR 1029; NIH DMID 02-184; Univ of Maryland IRB 0303311; HSRRB A-12093; NIAID IRB 177
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-05

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; malaria; merozoite surface protein-1
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- FMP1/AS02A Vaccine (Experimental): 500 uL of FMP1/AS02A is given to subject on days 0, 30+7, and 60+7 in the left deltoid muscle
  Interventions: Biological: FMP1/AS02A
- Imovax Rabies Vaccine (Active Comparator): 1 mL of Imovax Rabies Vaccine is given to subject on days 0, 30+7, and 60+7 in the left deltoid muscle
  Interventions: Biological: Imovax Rabies Vaccine

INTERVENTIONS:
Biological: FMP1/AS02A — FMP1 antigen contained 62.5 ug of lyophilized protein with 3.1 percent lactose as cryoprotectant. It's reconstituted in approx. 600 uL AS02A adjuvant manufactured by GSK. AS02A contains 50 ug MPL and 50ug QS21, 250uL of SB62 (oil/water emulsion) in phosphate buffered saline (PBS) per volume of 0.5 mL. All AS02A vials contained 0.65 to 0.75 mL of liquid.
  Arms: FMP1/AS02A Vaccine
Biological: Imovax Rabies Vaccine — Sterile, stable, freeze-dried suspension of rabies virus prepared from the strain PM-1503-3M, obtained from the Wistar Inst. in Philadelphia. Each 1 mL dose of vaccine contained 100 mg of human albumin, <150g of neomycin sulfate, and >2.5 IU of rabies antigen.
  Arms: Imovax Rabies Vaccine

SUMMARY:
This study tested the safety of a new malaria vaccine in adults in Mali, West Africa, and measured the ability of the vaccine to stimulate antibodies directed against the malaria protein that the vaccine is based on. Forty adults were randomly assigned to get either the experimental malaria vaccine or a rabies vaccine, for comparison.

DETAILED DESCRIPTION:
The study was a randomized, controlled trial in which participants and clinical investigators were blinded to vaccine group assignment. Forty adults were randomized in a 1:1 ratio to receive either FMP1/AS02A or the control rabies vaccine. The aims of the control group were to account for baseline morbidity and the impact of seasonal malaria transmission on the dynamics of anti-MSP-1 antibodies, and to minimize bias in assessment of adverse events. Vaccines were given on a 0-, 1- and 2-month schedule. The first immunization was given in early July just as malaria transmission began; the second dose at the end of July as transmission was increasing; and the third dose in late August near the peak of malaria transmission intensity. Study day 90 was in October, shortly after transmission crests and when severe and uncomplicated malaria disease episodes peak, study day 180 was at the end of the malaria season, and study day 272 was at the height of the dry season. The final study follow-up on day 364 coincided with the beginning of the 2004 malaria season. Interim safety analyses were reviewed by an independent Safety Monitoring Committee before the second and third immunizations.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant female aged 18-55 years inclusive at the time of screening.
* For women, willingness not to become pregnant until 1 month after the last dose of vaccine
* Written informed screening and study consent obtained from the participant before study start.
* Available and willing to participate in follow-up for the duration of study (12 months)

Exclusion Criteria:

* Previous vaccination with an investigational malaria vaccine or with any rabies vaccine.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose.
* Chronic administration (defined as more than 14 days) of immuno-suppressants or other immune-modifying drugs within six months prior to the first vaccine dose. This will include oral steroids and inhaled steroids, but not topical steroids.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of study vaccine(s) with the exception of tetanus toxoid.
* Previous vaccination with a vaccine containing MPL and/or QS-21 such as RTS,S.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Any confirmed or suspected autoimmune disease
* History of allergic reactions or anaphylaxis to immunizations or to any vaccine component.
* History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care
* History of allergy to tetracycline, doxycycline or neomycin
* History of splenectomy
* Serum ALT >=35 IU/L
* Serum creatinine level >133 micro moles per Liter (1.5 mg/dL)
* Hb <11 g/dL for males and <10 g/dL for females
* WBC <3.0 x 103/mm3 or >13.5 x 103/mm3
* Absolute lymphocyte count <=1.0 x 103 per micro liter
* Thrombocytopenia < 100,000 per micro liter
* More than trace protein, more than trace hemoglobin or positive glucose in urine
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Suspected or known current alcohol or illicit drug abuse.
* Pregnancy or positive urine beta-HCG on the day of or prior to immunization.
* Breastfeeding
* Simultaneous participation in any other interventional clinical trial.
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurologic condition, or any other findings that in the opinion of the PI may increase the risk to the participant from participating in the study.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-07; Primary Completion 2004-09 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou A Thera, MD MPH, Principal Investigator — University of Bamako Faculty of Medicine, Mali
Locations (1):
- Bandiagara Malaria Project, Bandiagara, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoute JA, Gombe J, Withers MR, Siangla J, McKinney D, Onyango M, Cummings JF, Milman J, Tucker K, Soisson L, Stewart VA, Lyon JA, Angov E, Leach A, Cohen J, Kester KE, Ockenhouse CF, Holland CA, Diggs CL, Wittes J, Heppner DG Jr; MSP-1 Malaria Vaccine Working Group. Phase 1 randomized double-blind safety and immunogenicity trial of Plasmodium falciparum malaria merozoite surface protein FMP1 vaccine, adjuvanted with AS02A, in adults in western Kenya. Vaccine. 2007 Jan 2;25(1):176-84. doi: 10.1016/j.vaccine.2005.11.037. Epub 2005 Dec 7. PMID 16388879
- [Background] Ockenhouse CF, Angov E, Kester KE, Diggs C, Soisson L, Cummings JF, Stewart AV, Palmer DR, Mahajan B, Krzych U, Tornieporth N, Delchambre M, Vanhandenhove M, Ofori-Anyinam O, Cohen J, Lyon JA, Heppner DG; MSP-1 Working Group. Phase I safety and immunogenicity trial of FMP1/AS02A, a Plasmodium falciparum MSP-1 asexual blood stage vaccine. Vaccine. 2006 Apr 5;24(15):3009-17. doi: 10.1016/j.vaccine.2005.11.028. Epub 2005 Nov 28. PMID 16356603
- [Derived] Thera MA, Doumbo OK, Coulibaly D, Diallo DA, Kone AK, Guindo AB, Traore K, Dicko A, Sagara I, Sissoko MS, Baby M, Sissoko M, Diarra I, Niangaly A, Dolo A, Daou M, Diawara SI, Heppner DG, Stewart VA, Angov E, Bergmann-Leitner ES, Lanar DE, Dutta S, Soisson L, Diggs CL, Leach A, Owusu A, Dubois MC, Cohen J, Nixon JN, Gregson A, Takala SL, Lyke KE, Plowe CV. Safety and immunogenicity of an AMA-1 malaria vaccine in Malian adults: results of a phase 1 randomized controlled trial. PLoS One. 2008 Jan 23;3(1):e1465. doi: 10.1371/journal.pone.0001465. PMID 18213374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 subjects were randomized at 1:1 ratio to receive either FMP1/AS02A or Imovax Rabies vaccine. All 40 subjects received all 3 immunizations and were followed for 12 months
Period: Overall Study
Arm/Group | FMP1/AS02A Vaccine | Imovax Rabies Vaccine
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMP1/AS02A Vaccine | Imovax Rabies Vaccine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (8.0) | 38.5 (10.0) | 39.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 15 | 18 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Mali | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events by Immunization and Type
Description: Number of participants with solicited adverse events by immunization and type (local, general and any) during each of the three eight-day follow-up periods after each vaccination (day of vaccination and post-vaccination days 1, 2, 3, and 7). Subjects were immunized on days 0, 30+7, and 60+7.
Time Frame: Days 0, 1, 2, 3, 7, 30, 31, 32, 33, 37, 60, 61, 62, 63, 67
Measure: Count of Participants; unit: Participants
Arm/Group | Imovax Rabies Vaccine | FMP1/AS02A Vaccine
Number analyzed (Participants) | 20 | 20
Participants
  Immunization 1: Any Symptom | 8 | 18
  Immunization 1: Local Symptom | 4 | 13
  Immunization 1: General Symptom | 4 | 14
  Immunization 2: Any Symptom | 12 | 13
  Immunization 2: Local Symptom | 7 | 10
  Immunization 2: General Symptom | 8 | 12
  Immunization 3: Any Symptom | 11 | 11
  Immunization 3: Local Symptom | 9 | 8
  Immunization 3: General Symptom | 5 | 8

2. Secondary Outcome: Geometric Mean Titers for Anti-FMP1 Antibody
Description: Immune response was measured by anti-FMP1 endpoint titers. Data were obtained on day 0, 14, 30, 44, 60, 74, 90, 180, 272, and 364. Samples collected on vaccination days (days 0, 30, and 60) were collected immediately prior to vaccination.
Time Frame: Days 0, 14, 30, 44, 60, 74, 90, 180, 272, and 364
Population: Immune response was measured by anti-FMP1 endpoint titers. Data were obtained on day 0, 14, 30, 44, 60, 74, 90, 180, 272, and 364. Samples collected on vaccination days (days 0, 30, and 60) were collected immediately prior to vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titers
Groups:
- Geometric Mean Titer: Geometric Mean Titer (GMT)
Arm/Group | Geometric Mean Titer
Number analyzed (Participants) | 40
geometric mean titers
  Imovax: Pre-Imm 1 | 3282 [1423 to 7568]
  Imovax: Imm 1+14 days | 3089 [1332 to 7161]
  Imovax: Pre-Imm 2 | 3485 [1391 to 8728]
  Imovax: Imm 2+14 days | 4036 [1796 to 9071]
  Imovax: Pre-Imm 3 | 6915 [3148 to 15190]
  Imovax: Imm 3+14 days | 7051 [3477 to 14300]
  Imovax: Imm 3+30 days | 6892 [3645 to 13029]
  Imovax: Day 180 | 9089 [3817 to 21645]
  Imovax: Day 272 | 6367 [2743 to 14779]
  Imovax: Day 364 | 5015 [2194 to 11462]
  FMP1/AS02A: Pre-Imm 1 | 5858 [2650 to 12950]
  FMP1/AS02A: Imm 1+14 days | 7627 [3561 to 16336]
  FMP1/AS02A: Pre-Imm 2 | 8007 [3809 to 16831]
  FMP1/AS02A: Imm 2+14 days | 20044 [12994 to 30919]
  FMP1/AS02A: Pre-Imm 3 | 26321 [19611 to 35326]
  FMP1/AS02A: Imm 3+14 days | 35194 [26245 to 47194]
  FMP1/AS02A: Imm 3+30 days | 37923 [26788 to 53686]
  FMP1/AS02A: Day 180 | 29150 [18301 to 46432]
  FMP1/AS02A: Day 272 | 19518 [11181 to 34072]
  FMP1/AS02A: Day 364 | 14693 [8216 to 26276]

ADVERSE EVENTS:
Time Frame: Solicited AEs were recorded during each of the 3 eight day follow-up periods after each vaccination and unsolicited AEs were recorded for 12 months
Description: Solicited AEs were recorded by occurrence of symptoms elicited during each of the three eight-day follow-up periods after each vaccination (day of vaccination and post-vaccination days 1, 2, 3, and 7). Subjects were immunized on days 0, 30+7, and 60+7. Unsolicited AEs were recorded for 12 months. AEs were listed by Vaccine group, per subject, and immunization number (1, 2, or 3).
  Grade 1= Easily tolerated; Grade 2= Interferes with daily activities; Grade 3= Prevents daily activities
Arm/Group | Imovax Rabies Vaccine | FMP1/AS02A Vaccine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/20
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imovax Rabies Vaccine (N=20) | FMP1/AS02A Vaccine (N=20)
Tubal ectopic pregnancy (right side) (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Immunization 3
Sinusitus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Immunization 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imovax Rabies Vaccine (N=20) | FMP1/AS02A Vaccine (N=20)
Arm motion limitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anus disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 1 (1) | 2 (2)
Ataxia (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bloody diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Bradypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chills (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8)
Chills (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 8 (8) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (3)
Fever (General disorders) | 3 (3) | 7 (7)
Fever (General disorders) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 5 (5) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 8 (8) | 20 (20)
Heart murmur (Cardiac disorders) | 1 (1) | 0 (0)
Hemorrhoids (Vascular disorders) | 0 (0) | 1 (1)
Hot flushes (Vascular disorders) | 10 (10) | 20 (20)
Infection (Infections and infestations) | 5 (5) | 10 (10)
Inflammation at injection site (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Lacrimation abnormal (Eye disorders) | 0 (0) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leukorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 3 (3) | 0 (0)
Malaise (General disorders) | 7 (7) | 8 (8)
Malaria (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Otitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pain at injection site (Injury, poisoning and procedural complications) | 6 (6) | 20 (20)
Pain at injection site (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pregnancy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus ocular (Eye disorders) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 8 (8) | 10 (10)
Rigors (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Saliva increased (Gastrointestinal disorders) | 1 (1) | 0 (0)
Site mass at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sweating increased (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 15 (15) | 20 (20)
Taste perversion (Nervous system disorders) | 1 (1) | 1 (1)
Thirst (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tooth ache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth caries aggrevated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vision accomodation abnormal (Eye disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No